CLINICAL TRIAL: NCT06784505
Title: Obstetric Outcomes of Primigravidae At Women's Health Centre; Cross Sectional Study
Brief Title: Obstetric Outcomes of Primigravidae
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menna Allah Abd Elaziaz Ahmed, Resident, Assiut University
Other Study IDs: Outcomes in primigravidae
Record Dates: First submitted 2025-01-10; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Primigravida Labour
Keywords: Primigravidae

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To determine obstetric outcomes in primigravida at term at women's health centre

DETAILED DESCRIPTION:
A primigravida is a woman carrying her first pregnancy(.1)A woman carrying her first pregnancy is starting a new life and it is a crucial time in her obstetric career as subsequent obstetric performance will depend on how well the first pregnancy was managed.(2).Pregnancy in a primigravida is often viewed with anxiety not only by the patient who is going through the experience for the first time but also her relatives and her caregiver. The obstetric outcome of primigravidae is associated with many complications; therefore, they are considered high risk because of both maternal and fetal concerns(.2).Numerous studies have shown that primigravidae are at increased risk of complications during pregnancy, labor, and delivery and if not properly managed, these complications can result in increased morbidity and mortality for both the mother and baby(3) Reported complications include abnormal labor patterns, increased risk of operative deliveries, increased rate of admissions into neonatal intensive care unit and increased perinatal deaths.(4,5,6) The cardinal observation to be made in a gravid uterus at term in labor is engagement of head which is the initial step in the mechanism of labor. The term "engagement" in normal labor denotes that the greatest diameter of fetal head has passed through the brim of the pelvis.(7) Engaged head in a primigravida at term in early labor is a sign of pelvic adequacy.Unengaged head at the onset of labor is associated with increase in duration of labor and incidence of dysfunctional labor pattern.(8,9) Thus, undue prolongation of labor leads to increased risk of caesarean section(10,11) and its associated maternal and perinatal morbidity and mortality. The adequacy of the pelvis, the efficacy of uterine contractions, the capacity of fetal head to mold and the temperamental resilience of the patient contribute more to the outcome of labor. Hence, the dynamics of labor is equally important with mechanics as it improves the adaptation of fetal head To the pelvic cavity and its passage through it supported by primary and secondary forces of labor. Careful monitoring of progress of labor and timely medical intervention in these cases can reduce the incidence of caesarean deliveries. (11)This study will, therefore, assess the obstetric outcome of vaginal delivery of these women at term considering course & duration of labour & the incidence of complication with its associated fetomaternal outcomes

ELIGIBILITY:
Inclusion Criteria:

* Primigravida with singleton live fetus
* Cephalic presentation
* Delivered at term with gestational age(37 -41 weeks)

Exclusion Criteria:

* Multiparous women
* Multiple gestation
* Intra Uterine fetal death th (IUFD)
* Medical condition as preclampsia
* Polyhydramnios and fetal anomalies
* Malpresentation (e.g., breech, face).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primigravida in labor satisfying the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Maternal outcome | 10 hours
  Maternal outcome woth respect to course of labour & duration of first and second stage of labour

SECONDARY OUTCOMES:
Progress of labour & neonatal outcome | 10 hours
  Progress of labour in the respect of needing augmentation,mode of delivery & labour complications Neonatal outcome in the respect of Apgar score, birth weight & NICU admissions

REFERENCES:
- See also: Arti Kumari1,Anupama Sinha2.(2024)A Feto-Maternal Outcome of Primigravida with Unengaged Head at Term.International Journal of Pharmaceutical and Clinical Research ; 16(7); 998-1002 — https://www.ijrcog.org/index.php/ijrcog/article/view/14616
- See also: L., R., Sujatha Prabhu, & Kusuma Naik M. V. (2023). Maternal and fetal outcome in primigravida with unengaged head at term in labour. International Journal of Reproduction, Contraception, Obstetrics and Gynecology, 12(6), 1569-1574. — https://www.ijrcog.org/index.php/ijrcog/article/view/12981
- See also: Priya Agarwal, Shraddha Shetty. Clinical study of primigravida with unengaged head in labour at term .Int J Women's Health Rerpod Sci 9, 2021 — https://www.researchgate.net/publication/348642844_Clinical_Study_of_Primigravida_With_Unengaged_Head_in_Labour_at_Term
- See also: Orji EO, Ndububa VI. Obstetric performance of women aged over forty years. East Afr Med J. 2004;81:139-41. doi: 10.4314/eamj.v81i3.9143. [DOI] [PubMed] [Google Scholar] — https://pubmed.ncbi.nlm.nih.gov/15293972/
- See also: Ogedengbe OK, Odeneye TO. Outcome of Instrumental deliveries in Lagos Nigeria. Implications for its use at the second tier healthcare level. Nig Med Pract. 2006;45:106-10. [Google Scholar] — https://www.researchgate.net/publication/315089308_Outcome_of_Instrumental_Deliveries_in_Lagos_Nigeria_Implications_For_its_Use_at_the_Second_Tier_Healthcare_Level
- See also: .Danish N, Fawad A, Abbasi N. Assessment of pregnancy outcome in primigravida: Comparison between booked and un-booked patients. J Ayub Med Coll Abbottabad. 2010;22:23-5. [PubMed] [Google Scholar] — https://pubmed.ncbi.nlm.nih.gov/21702258/